CLINICAL TRIAL: NCT05246332
Title: Grounding the Body Improves Sleep Quality in Patients With Mild Alzheimer's Disease
Brief Title: Grounding Effect on Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 201901136B0
Record Dates: First submitted 2022-02-09; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2019-08

CONDITIONS: Alzheimer Disease; Insomnia; Depression, Anxiety
MeSH Terms: conditions — Alzheimer Disease; Sleep Initiation and Maintenance Disorders; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The investigators use a grounding wire and a sham grounding wire to create grounding and sham-grounding groups. The patients are blinded to the grounding because they do not know which one has a grounding effect according to the exterior of the mat.
  The investigators who do the evaluation of questionnaire and electrochemical analyzer and the outcomes assessor who interpret the data do not know which wire has grounding effect, too.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient receive grounding (Experimental): The investigators use the grounding mat (EARTHING Conductive Earthing Uni-versal Mat with Earthing Cord) as the grounding method. The grounding group use a grounding wire to sit on a chair barefoot in contact with the grounding mat for 30 minutes.
  Interventions: Device: Grounding
- Patient receive sham-grounding (Sham Comparator): The investigators use the grounding mat (EARTHING Conductive Earthing Uni-versal Mat with Earthing Cord) as the grounding method. The sham-grounding group use a sham grounding wire to sit on a chair barefoot in contact with the grounding mat for 30 minutes.
  Interventions: Device: Grounding

INTERVENTIONS:
Device: Grounding — The investigators used a grounding wire and a sham grounding wire to create grounding and sham-grounding groups. Participants sat on a chair barefoot in contact with the grounding mat for 30 minutes. The participants were blinded to the grounding because they did not know which one had a grounding effect according to the exterior of the mat.

SUMMARY:
The investigators explore the effectiveness of grounding as a non-pharmacological therapy for treating sleep disturbances, anxiety, and depression in patients with mild AD.

DETAILED DESCRIPTION:
Grounding refers to having direct contact with the Earth, such as walking barefoot or lying on the ground. Research has found that grounding can improve inflammation, free radical damage, blood pressure, sleep quality, pain, stress, mood, and wound healing. However, there has been no re-search on the effect of utilizing grounding for patients with Alzheimer's disease (AD). Thus, in this study, the investigators explore the effectiveness of grounding as a non-pharmacological therapy for treating sleep disturbances, anxiety, and depression in patients with mild AD.

Patients with mild AD were enrolled in the study. The electrochemical analyzer CHI 1205b was employed to check the electrochemical signals at acupoints KI1 and GV16. The investigators used the Pittsburgh Sleep Quality Index (PSQI), Beck Anxiety Inventory (BAI), and Beck Depression Inventory-II (BDI-II) to evaluate sleep quality, anxiety, and depression, respectively, at weeks 0 and 12.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with dementia, and CDR ≥ 0.5
* aged > 50 years,
* sit with bilateral bare feet on the grounding mat
* able to answer the questionnaire
* able to sign the informed consent adequately.

Exclusion Criteria:

* aged less than 50 years
* inability to sit with bilateral bare feet on the grounding mat
* currently taking anti-oxidative health supplements or anti-inflammatory medicine.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
The Pittsburgh Sleep Quality Index (PSQI) questionnaire for insomnia, score range from 0 to 21, the higher score means worse sleep quality | through study completion, an average of 12 weeks.
  The investigators measure Pittsburgh Sleep Quality Index (PSQI) score before the patients participate the study (week 0, baseline data). After receiving 12 weeks grounding, the investigators measure PSQI again (week 12, post grounding data).
The Beck Anxiety Inventory (BAI) questionnaire for anxiety, score range from 0 to 63, the higher score means more anxiety the patient is. | through study completion, an average of 12 weeks.
  The investigators measure Beck Anxiety Inventory (BAI) score before the patients participate the study (week 0, baseline data). After receiving 12 weeks grounding, the investigators measure BAI again (week 12, post grounding data).
The Beck Depression Inventory-II (BDI-II) questionnaire for depression, score range from 0 to 63, the higher score means more depression the patient is. | through study completion, an average of 12 weeks.
  The investigators measure Beck Depression Inventory-II (BDI-II) score before the patients participate the study (week 0, baseline data). After receiving 12 weeks grounding, the investigators measure BDI-II again (week 12, post grounding data).
The electric current | through study completion, an average of 12 weeks.
  The electrochemical analyzer CHI 1205b is a device that can measure the electric current via reduction-oxidation reaction.
  The investigators measure the electric current before the patients participate the study (week 0, baseline data). After receiving 12 weeks grounding, the investigators measure the electric current again (week 12, post grounding data).

CONTACTS AND LOCATIONS:
Overall Officials: Nai-Ching Chen, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Menigoz W, Latz TT, Ely RA, Kamei C, Melvin G, Sinatra D. Integrative and lifestyle medicine strategies should include Earthing (grounding): Review of research evidence and clinical observations. Explore (NY). 2020 May-Jun;16(3):152-160. doi: 10.1016/j.explore.2019.10.005. Epub 2019 Nov 14. PMID 31831261
- [Background] Figueiro MG, Plitnick B, Roohan C, Sahin L, Kalsher M, Rea MS. Effects of a Tailored Lighting Intervention on Sleep Quality, Rest-Activity, Mood, and Behavior in Older Adults With Alzheimer Disease and Related Dementias: A Randomized Clinical Trial. J Clin Sleep Med. 2019 Dec 15;15(12):1757-1767. doi: 10.5664/jcsm.8078. Epub 2019 Nov 8. PMID 31855161
- [Background] Whitney MS, Shemery AM, Yaw AM, Donovan LJ, Glass JD, Deneris ES. Adult Brain Serotonin Deficiency Causes Hyperactivity, Circadian Disruption, and Elimination of Siestas. J Neurosci. 2016 Sep 21;36(38):9828-42. doi: 10.1523/JNEUROSCI.1469-16.2016. PMID 27656022